CLINICAL TRIAL: NCT06457438
Title: Molecular Characteristics and Prevalence of Viral Hepatitis E in Human Tissue and Cell Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05/OR-FNOs/2024; 05/OR-FNOs/2024 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis E
Keywords: Hepatitis E; Organ Donor; Cell Donor; HEV RNA
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Intervention Model Description: The study subjects and their samples will be divided into two study groups.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organ Donors (Experimental): Samples obtained from organ donors will be included in this study arm.
  Interventions: Diagnostic Test: Elecsys Anti-HEV IgG, IgM
- Cell Donors (Experimental): Samples obtained from cell donors will be included in this study arm.
  Interventions: Diagnostic Test: Elecsys Anti-HEV IgG, IgM

INTERVENTIONS:
Diagnostic Test: Elecsys Anti-HEV IgG, IgM — Diagnostic test used to determine antibodies in blood and serum.

SUMMARY:
In this study, the researchers want to focus on the prevalence of anti-HEV antibodies by a new generation test, direct detection of HEV RNA, and its genotypic analysis in a group of human tissue and cell donors.

DETAILED DESCRIPTION:
At the Department of Laboratory Medicine of the Faculty of Medicine of the Faculty of Medicine of the National University of Health Sciences, human tissue and cells from donors will be examined for the assessment of health eligibility and donor selection according to Decree No. 422/2008 Coll. According to the current legislation, the determination of IgG and IgM antibodies against HEV or the HEV RNA method is not part of the standard examination of human tissue and cell donors for the assessment of their health eligibility.

ELIGIBILITY:
Inclusion Criteria:

- patients indicated for organ or cell donation

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hepatitis E in the study groups | 2 years
  The prevalence of Hepatitis E will be observed in both study groups, measured as the number of positive samples from the total number of samples.

SECONDARY OUTCOMES:
Presence of Hepatitis E (HEV) RNA in the study groups | 2 years
  The presence of HEV RNA will be observed in both study groups, measured as the number of positive samples from the total number of samples.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Slepčanová, Mgr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Tedder RS, Ijaz S, Kitchen A, Ushiro-Lumb I, Tettmar KI, Hewitt P, Andrews N. Hepatitis E risks: pigs or blood-that is the question. Transfusion. 2017 Feb;57(2):267-272. doi: 10.1111/trf.13976. PMID 28194857
- [Background] Horvatits T, Schulze Zur Wiesch J, Lutgehetmann M, Lohse AW, Pischke S. The Clinical Perspective on Hepatitis E. Viruses. 2019 Jul 5;11(7):617. doi: 10.3390/v11070617. PMID 31284447
- [Background] Kamar N, Izopet J, Pavio N, Aggarwal R, Labrique A, Wedemeyer H, Dalton HR. Hepatitis E virus infection. Nat Rev Dis Primers. 2017 Nov 16;3:17086. doi: 10.1038/nrdp.2017.86. PMID 29154369
- [Background] Blasco-Perrin H, Madden RG, Stanley A, Crossan C, Hunter JG, Vine L, Lane K, Devooght-Johnson N, Mclaughlin C, Petrik J, Stableforth B, Hussaini H, Phillips M, Mansuy JM, Forrest E, Izopet J, Blatchford O, Scobie L, Peron JM, Dalton HR. Hepatitis E virus in patients with decompensated chronic liver disease: a prospective UK/French study. Aliment Pharmacol Ther. 2015 Sep;42(5):574-81. doi: 10.1111/apt.13309. Epub 2015 Jul 14. PMID 26174470
- [Background] Kumar A, Saraswat VA. Hepatitis E and Acute-on-Chronic Liver Failure. J Clin Exp Hepatol. 2013 Sep;3(3):225-30. doi: 10.1016/j.jceh.2013.08.013. Epub 2013 Sep 16. PMID 25755504
- [Background] Nemecek V, Butovicova P, Maly M, Dite P, Vertatova M, Vodickova I, Kriz B. [The prevalence of antibodies against Hepatitis E Virus in the Czech Republic: serological survey]. Epidemiol Mikrobiol Imunol. 2017 Winter;66(1):3-7. Czech. PMID 28374592
- See also: World Health Organization. Hepatitis E: Fact sheet — https://www.who.int/en/news-room/fact-sheets/detail/hepatitis-e